CLINICAL TRIAL: NCT01018628
Title: A Phase I Randomized, Placebo-Controlled, Single-Blind, Multiple-Dose, Dose-Escalation Clinical Study to Assess the Safety and Pharmacokinetics of SRT2379 in Normal Healthy Male Volunteers
Brief Title: A Clinical Study to Assess the Safety and Pharmacokinetics of SRT2379 in Normal Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 114011
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 - Dose Level A (25 mg/day) (Active Comparator): Cohort 1 will be administered at approximately the same time every dosing day after fasting for 10hrs. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving 25 mg SRT2379 and one subject receiving placebo. The remainder of subjects in this cohort will be dosed on Day 2 of the single dose period with five subjects receiving 25 mg SRT2379 and one subject receiving placebo, assuming that no significant safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study. The other cohorts will be dosed sequentially allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort.
  Interventions: Drug: SRT2379; Drug: Placebo
- Cohort 2 - Dose Level B (75 mg/day) (Active Comparator): Cohort 2 will be administered at approximately the same time every dosing day after fasting for 10hrs. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving 75 mg SRT2379 and one subject receiving placebo. The remainder of subjects in this cohort will be dosed on Day 2 of the single dose period with five subjects receiving 75 mg SRT2379 and one subject receiving placebo, assuming that no significant safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study. The other cohorts will be dosed sequentially allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort.
  Interventions: Drug: SRT2379; Drug: Placebo
- Cohort 3 - Dose Level C (250 mg/day) (Active Comparator): Cohort 3 will be administered at approximately the same time every dosing day after fasting for 10hrs. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving 250 mg SRT2379 and one subject receiving placebo. The remainder of subjects in this cohort will be dosed on Day 2 of the single dose period with five subjects receiving 250 mg SRT2379 and one subject receiving placebo, assuming that no significant safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study. The other cohorts will be dosed sequentially allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort.
  Interventions: Drug: SRT2379; Drug: Placebo
- Cohort 4 - Dose Level D (500 mg/day) (Active Comparator): Cohort 4 will be administered at approximately the same time every dosing day after fasting for 10hrs. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving 500 mg SRT2379 and one subject receiving placebo. The remainder of subjects in this cohort will be dosed on Day 2 of the single dose period with five subjects receiving 500 mg SRT2379 and one subject receiving placebo, assuming that no significant safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study. The other cohorts will be dosed sequentially allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort.
  Interventions: Drug: SRT2379; Drug: Placebo
- Cohort 5 - Dose Level E (1000 mg/day) (Active Comparator): Cohort 5 will be administered at approximately the same time every dosing day after fasting for 10hrs. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving 1000 mg SRT2379 and one subject receiving placebo. The remainder of subjects in this cohort will be dosed on Day 2 of the single dose period with five subjects receiving 1000 mg SRT2379 and one subject receiving placebo, assuming that no significant safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study. The other cohorts will be dosed sequentially allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort.
  Interventions: Drug: SRT2379; Drug: Placebo
- Cohort 6 - Dose Level F (2000 mg/day) (Active Comparator): Cohort 6 will be administered at approximately the same time every dosing day after fasting for 10hrs. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving 2000 mg SRT2379 and one subject receiving placebo. The remainder of subjects in this cohort will be dosed on Day 2 of the single dose period with five subjects receiving 2000 mg SRT2379 and one subject receiving placebo, assuming that no significant safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study. The other cohorts will be dosed sequentially allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort.
  Interventions: Drug: SRT2379; Drug: Placebo
- Cohort 7 - Dose Level G (3000 mg/day) (Active Comparator): Cohort 7 will be administered at approximately the same time every dosing day after fasting for 10hrs. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving 3000 mg SRT2379 and one subject receiving placebo. The remainder of subjects in this cohort will be dosed on Day 2 of the single dose period with five subjects receiving 3000 mg SRT2379 and one subject receiving placebo, assuming that no significant safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study. The other cohorts will be dosed sequentially allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort.
  Interventions: Drug: SRT2379; Drug: Placebo
- Cohort 8 - Dose Level H (500 mg/day in fed state) (Active Comparator): Cohort 8 will be administered at approximately the same time every dosing day and 30 minutes following the start of consumption of a standardized high-fat meal. Two subjects will be dosed on Day 1 of the single dose period with one subject receiving SRT2379 and one subject receiving placebo. The remainder of subjects in this cohort will be dosed on Day 2 of the single dose period with five subjects receiving SRT2379 and one subject receiving placebo, assuming that no significant safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study. The dose of SRT2379 administered to subjects in the fed state is planned to be 500 mg, however this may be modified upwards or downwards following evaluation of safety and pharmacokinetic data from earlier cohorts. The fed cohort will be the final cohort dosed in the study.
  Interventions: Drug: SRT2379; Drug: Placebo

INTERVENTIONS:
Drug: SRT2379 — SRT2379 will be supplied as hard gelatin capsules, with each containing 25 mg or 250 mg of SRT2379 free base equivalent (31 or 310 mg of SRT2379 monosuccinate) without any additive.
Drug: Placebo — For placebo product, the SRT2379 drug substance will be replaced by Microcrystalline Cellulose (Avicel® PH 200) to match the SRT2379 investigational product.

SUMMARY:
The main purpose of this study is to assess the safety and pharmacokinetics of SRT2379 (25, 75, 250, 500, 1000, 2000, and 3000 mg/day [fasted] and 500 mg/day [fed]) in healthy male volunteers.

The purpose is also to explore the effect of SRT2379 on plasma concentrations of Fibroblast Growth Factor 21 (FGF21) and to identify other possible biomarkers suitable for future clinical assessment of oral SIRT1 activators.

DETAILED DESCRIPTION:
Prospective, single center, clinical study of SRT2379 administered orally. Randomized, placebo-controlled, single-blind, multiple-dose, dose-escalation inpatient/outpatient study to assess the safety and pharmacokinetics (PK) of SRT2379 in healthy male volunteers. Approximately sixty-four (64) subjects aged 18-55, who fulfill the inclusion/exclusion criteria, will be enrolled in this study. Eight cohorts of eight subjects each will be examined. Subjects within each cohort will be randomized 6:2 to receive SRT2379 at one of seven escalating doses (A, B, C, D, E, F or G), likely to be 25, 75, 250, 500, 1000, 2000, and 3000 mg/day or placebo. All cohorts will be administered SRT2379 in the fasted state, with the exception of one cohort that will receive one of the stated doses of SRT2379 in the fed state (the dose of SRT2379 administered to subjects in the fed state is planned to be 500 mg, however this may be modified upwards or downwards following evaluation of safety and pharmacokinetic data from earlier cohorts. The fed cohort will be the final cohort dosed in the study.). Two subjects will be dosed on Day 1 of the single dose period with one subject receiving active treatment and one subject receiving placebo. The remainder of subjects within each cohort will be dosed on Day 2 of the single dose period with five subjects receiving active treatment and one subject receiving placebo, assuming that no safety issues arise in the two subjects dosed on Day 1. Subjects will remain on a fixed dose of test material for all dosing days in the study.

Each cohort of subjects will be dosed sequentially approximately three weeks apart for the single dose period, and return to the study unit approximately two weeks after their single dose administration to receive 7 consecutive days of dosing for the multiple-dose period. Each cohort of subjects in the multiple-dose period will be dosed sequentially, approximately, two weeks apart (from multiple dose period Day 7 of preceding cohort to multiple dose period Day 1 dose of the subsequent cohort), allowing for a comprehensive safety assessment prior to initiation of an escalated dose in a subsequent cohort.

Subjects will sign the informed consent form at the Screening Visit. If eligible and willing to participate, subjects will enter into the study. Subjects will have fasted for at least 10 hours overnight and be randomized to receive SRT2379 or placebo (test material). The subject cohort assigned to the fed dose will consume a standardized meal before receiving test material; all other subjects will receive test material in a fasted state. Subjects will be required to stay overnight at the study unit for two nights during the single dose period of the study and subsequently, for the duration of the seven-day multiple-dose period (8 consecutive overnight stays) to assess safety and to gather required PK samples. Subjects will be asked to return to the study center for an End of Study safety assessment approximately 1 week after the last administration of study drug during the multiple-dose period.

Dose escalation will be dependent on safety parameters (physical examination findings, vital signs, ECG studies, adverse events and laboratory values) and PK data.

ELIGIBILITY:
Inclusion Criteria:

* Be male within the age range of 18 to 55 years.
* Voluntarily sign an Independent Review Board/Research Ethics Committee (IRB/REC)-approved informed consent form to participate in the study after all relevant aspects of the study have been explained and discussed with the subject.
* Have Hematology, Coagulation, Clinical Chemistry and Urinalysis test results that are within normal, allowable limits (if out-of-range, must be considered clinically significant by the Principal Investigator to be exclusionary) and performed within 21 days of receiving first dose of test material. In addition, the Principal Investigator will discuss any out-of-range electrolyte values with Sirtris' medical monitor for assessment of clinical significance.
* Have a BMI (Body Mass Index) ≥18.0 and ≤30.0 kg/m^2.
* Be clear of any history of HIV 1 and 2 and hepatitis B and C.
* Have no significant disease or clinically significant abnormal laboratory value as deemed by the Investigator on the laboratory evaluations, medical history, or physical exam.
* Have a normal 12-lead ECG or an ECG with abnormality considered to be clinically insignificant. Specifically, the QTcB must be ≤ 450 msec, and no evidence of bundle branch block must be present.
* Have the ability to communicate with the investigative site staff in a manner sufficient to carry out all protocol procedures as described.
* Subject and his partner must agree to use an acceptable double barrier method for birth control from the Screening visit through 3 months after the last dose of test material.

Exclusion Criteria:

* Subject has had a major illness in the past three months or any significant ongoing chronic medical illness that the Investigator would deem unfavorable for enrollment.
* Subject has renal or liver impairment.
* Subject has clinically significant findings on Screening 24 hour 12-lead Holter.
* Subject has a history of gastro-intestinal surgery or has a current gastrointestinal disease which may influence drug absorption.
* Subject has a history, within 3 years, of drug abuse (including benzodiazepines, opioids, amphetamine, cocaine, and THC) or a positive drug result at Screening.
* Subject has a history of smoking, within 3 months, or is currently a smoker.
* Subject has a history of alcoholism, and/or is currently drinking more than three drinks per day on a regular basis [one drink is equal to one unit of alcohol (one glass of wine, half a pint of beer, one measure of a spirit)].
* Subject has participated in a clinical trial within the past three months.
* Subject has a history of difficulty in donating blood or accessibility of veins in left or right arm.
* Subject has donated blood (one unit or 350 mL) within three months prior to receiving test material.
* Subject is taking herbal and dietary supplements or prescription drug therapy for which 5 times the half-life is longer than 21 days (i.e., the Screening period) prior to enrollment into the study. Please note: subjects must refrain from taking herbal or dietary supplements for the duration of the study.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-12-07 (Actual); Primary Completion 2010-08-06 (Actual); Study Completion 2010-08-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of SRT2379 (25, 75, 250, 500, 1000, 2000, 3000 mg/day [fasted] and 500 mg/day [fed]) in healthy male volunteers after single and multiple dose administration in the fasted and fed states. | Single Dose Period PK samples will be collected on Day1 at 0h, 15min, 30min, 1, 2, 4, 8, 12 and 24hrs post-dose. Multiple Dose Period PK samples will be collected on Days1-6 at 0h only, and on Day7 at 0h, 15min, 30min, 1, 2, 4, 8, 12 and 24hrs post-dose.
To determine the pharmacokinetic profile of SRT2379 (25, 75, 250, 500, 1000, 2000, 3000 mg/day [fasted] and 500 mg/day [fed]) in healthy male volunteers after single and multiple dose administration in the fasted and fed states. | AEs and clinically significant abnormal lab values will be recorded based upon Investigator observation and subject reporting. Safety will be monitored by AEs, VS, physical exam, labs and ECGs during the study.

SECONDARY OUTCOMES:
To explore the effect of SRT2379 (25, 75, 250, 500, 1000, 2000, and 3000 mg/day [fasted] and 500 mg/day [fed]) on plasma concentrations of Fibroblast Growth Factor 21 (FGF21). | Biomarker samples for plasma FGF-21 analysis will be collected on Day1 (single dose period) and Day7 (multiple dose period) at 0h, 1h, 4h, 8h post-dose and 24hrs post-dose on Days2 (single dose period) and 8 (multiple dose period).
To identify other possible biomarkers suitable for future clinical assessment of oral SIRT1 activators. | Blood samples for analysis of exploratory biomarkers will be collected on Day1 (single dose period) and Day7 (multiple dose period) at 0h, 1h, 4h, 8h post-dose and 24hrs post-dose on Days2 (single dose period) and 8 (multiple dose period).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Merthyr Tydfill, Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] GSK has concluded that it is not feasible to publish this study in a peer-reviewed scientific journal because the nature of the study is unlikely to be of interest to a journal. GSK is providing a results summary with a conclusion.
- See also: Results for study 114011 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114011?search=study&study_ids=114011#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register